CLINICAL TRIAL: NCT05876663
Title: Effect of Kinesio Taping on Pulmonary Function and Forward Shoulder Posture of Young Adults
Brief Title: Effect of Kinesio Taping on Pulmonary Function and Forward Shoulder Posture FSP of Young Adults
Acronym: FSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Saba Khan
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Healthy Young Adults
Keywords: Forward Shoulder Posture; Pulmonary Function; Kinesio Taping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping along with conventional physiotherapy protocol (Experimental): All baseline measurements will be collected in the beginning. In participant of experimental group the K-tape will be first applied from the anterior aspect of the acromion process of the scapular to the spinous process of the fourth thoracic vertebra (T4). Then, the K-tape will be applied from same origin to the insertion at the spinous process of the tenth thoracic vertebra (T10). K-tape will be applied with 50% tension of its original length.
  The K-tapes will be replaced with new ones every two days for six weeks. The outcome measures will be assessed after every two weeks i.e. pre-assessment, on week 2, week 4, and week 6.
  Primary outcome measures include the effect of kinesio taping on pulmonary function (via Digital Spirometry) and chest expansion (via Measuring Tape).Secondary outcome measures include FSP and pectoralis minor index (via Digital Vernier Caliper)
  Interventions: Other: Kinesio Taping; Other: Conventional physiotherapy protocol
- Conventional physiotherapy protocol (Active Comparator): Stretching exercise for Pectoralis Minor and Major muscle: Participant in supine lying try to touch the tip of shoulder with the bed surface e.g. retraction. Than in supine raise/abduct the arm at 90 and 120 degrees; try to drop down from the surface of the bed. Hold for 10 seconds 10 reps. 2 sessions per day for 6 weeks.
  Strengthening of Rhomboids: Participant in sitting position instructed to depress and retract the shoulder at the same time .Hold for 20 seconds 10 reps. 2 sessions per day for 6 weeks.
  Strengthening of lower and mid trapezius: In prone lying abduct arms to the side 90 degrees. Raise arms form surface of bed like an aero plane wings. Take a weight of 1 kg in hands and hold for 10 sec and 10 reps. 2 sessions per day for 6 weeks.
  Deep Breathing exercise: participant instructed to take a slow and deep breath inhaling through nose and exhaling through mouth. 10 rep 3 sessions per day for 6 weeks.
  Education regarding posture correction.
  Interventions: Other: Conventional physiotherapy protocol

INTERVENTIONS:
Other: Kinesio Taping — Kinesio Taping will be applied for 6 weeks and it will be changed with new one after every two days
  Arms: Kinesio Taping along with conventional physiotherapy protocol
Other: Conventional physiotherapy protocol — Stretching exercise for pectoralis minor and major:10 sets and 2 sessions per day for 6 weeks.
  Strengthening of Rhomboids and Trapezius muscle: 10 sets and 2 sessions per day for 6 weeks.
  Deep Breathing: 10 rep and 2 sessions per day for 6 weeks.

SUMMARY:
The aim of the study is to evaluate the effect of kinesio taping on pulmonary function and forward shoulder posture in young adults. Limited literature shows an association between forward shoulder posture and pulmonary function but the effect of kinesio taping for correction of forward shoulder posture and its consequences on pulmonary function is lacking in previous studies.

DETAILED DESCRIPTION:
Electronic devices and gadgets are mostly used for official and personal needs in this modern era. This increased usage leads to poor posture, especially in young adults. The FSP is the most common incorrect posture in youngsters. A study on posture correction shows the prevalence of rounded shoulders is 84% in the young adult age group of (18 to 24 years). The misaligned posture causes changes in anatomical structure leading to many musculoskeletal problems. Along with the musculoskeletal system, FSP also decreases chest wall mobility, lung capacities, and overall respiratory function. The respiratory muscle's proper functions is need to expand the thoracic cavity . The pectoralis muscles function is to elevate the rib cage and its tightness leads to lower chest expansion. Rhomboids play a role in stabilizing the scapula which helps the serratus muscle in forced inspiration. Weakness of middle and lower trapezius muscles causes the inability to straighten the back, thus affecting the ability to raise and expand the chest properly. Currently, for posture correction, usually in the form of conservative treatments such as stretching and strengthening exercises, McKenzie's exercises, Pilates, shoulder support braces, electrical modalities, etc are used to correct or reduce FSP. It is a dire need to find out the best physiotherapy approach for the correction of forward shoulder posture as well as improvement in pulmonary function that is not time-consuming like other exercise interventions. If the effectiveness of kinesio taping on pulmonary function is verified it will contribute to future use as the most suitable and less time-consuming approach in youngsters with FSP.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants
* Age: 18 - 25 years
* BMI within the normal range (18.5 to 24.9)
* Healthy participants with FSP

Exclusion Criteria:

* Skin allergies to elastic tape
* Known case of smokers
* Known cases of cardiovascular and pulmonary problems.
* Subjects with musculoskeletal disorders
* History of chronic neck or shoulder pain (NPRS >3)
* Any deformities or any condition that make it difficult to apply the Kinesio-Tape
* Those who refuse to participate
* Previous experience in respiratory muscle training

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | After 6 weeks
  Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings
Forced vital capacity (FVC) | After 6 weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
  Changes in FVC from baseline to 5th and after 15th day of intervention will be assessed.
Forced expiratory volume in 1sec (FEV1) | After 6 weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
Chest Expansion | After 6 weeks
  Chest expansion is the difference in thoracic girth after maximum inspiration and maximum expiration, which is one indicator of chest wall mobility. As it is measured using a measuring tape, it is a simple, inexpensive, and noninvasive tool for assessing chest mobility.

SECONDARY OUTCOMES:
Forward Shoulder Posture | After 6 weeks
  The forward shoulder posture (FSP) is characterized by downward rotation and anterior tilt of the scapula
Pectoralis Minor Index | After 6 weeks
  Pectoralis Minor Index (PMI) is a proposed parameter to evaluate the pectoralis minor length (PML), eliminating the effect of subject's variability of height.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Northwest Institute of Health Sciences, Peshawar, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MS, Cha YJ, Choi JD. Correlation between forward head posture, respiratory functions, and respiratory accessory muscles in young adults. J Back Musculoskelet Rehabil. 2017 Aug 3;30(4):711-715. doi: 10.3233/BMR-140253. PMID 28453447
- [Background] Carvalho LACM, Aquino CF, Souza TR, Anjos MTS, Lima DBM, Fonseca ST. Clinical Measures Related to Forward Shoulder Posture: A Reliability and Correlational Study. J Manipulative Physiol Ther. 2019 Feb;42(2):141-147. doi: 10.1016/j.jmpt.2019.03.006. Epub 2019 Apr 15. PMID 31000344
- [Background] Fani M, Ebrahimi S, Ghanbari A. Evaluation of scapular mobilization and comparison to pectoralis minor stretching in individuals with rounded shoulder posture: A randomized controlled trial. J Bodyw Mov Ther. 2020 Oct;24(4):367-372. doi: 10.1016/j.jbmt.2020.07.021. Epub 2020 Jul 30. PMID 33218535
- [Background] Shih HS, Chen SS, Cheng SC, Chang HW, Wu PR, Yang JS, Lee YS, Tsou JY. Effects of Kinesio taping and exercise on forward head posture. J Back Musculoskelet Rehabil. 2017;30(4):725-733. doi: 10.3233/BMR-150346. PMID 28282792
- [Background] Tomruk M, Keles E, Ozalevli S, Alpaydin AO. Effects of thoracic kinesio taping on pulmonary functions, respiratory muscle strength and functional capacity in patients with chronic obstructive pulmonary disease: A randomized controlled trial. Explore (NY). 2020 Sep-Oct;16(5):332-338. doi: 10.1016/j.explore.2019.08.018. Epub 2019 Sep 18. PMID 31611155